CLINICAL TRIAL: NCT00343278
Title: Post-Marketing Clinical Study of Valaciclovir Hydrochloride Tablets -Single Oral Dose Study in Hemodialysis Patients-
Brief Title: Pharmacokinetic Study Of Valaciclovir Hydrochloride Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104689
Record Dates: First submitted 2006-06-21; First posted 2006-06-22 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Virus Diseases
Keywords: Valaciclovir Hydrochloride; hemodialysis patient; ALDH; pharmacokinetics; Japanese
MeSH Terms: conditions — Virus Diseases | interventions — Valacyclovir

INTERVENTIONS:
Drug: Valaciclovir Hydrochloride

SUMMARY:
Valaciclovir (VACV), the L-valyl ester prodrug of aciclovir (ACV), is extensively converted to ACV and L-valine after oral administration. In subjects with normal renal function, ACV is predominantly eliminated unchanged in the urine, with a small proportion metabolized to 9-carboxymethoxymethylguanine (CMMG). The metabolism of ACV to CMMG is thought to involve aldehyde dehydrogenase (ALDH). On the basis of a high proportion of the Japanese population having low-activity ALDH, it can be hypothesized that the conversion of ACV to CMMG is decreased, thereby leading, in patients with renal impairment, to higher plasma concentrations of ACV. This pilot study was conducted to investigate potential relationships between genetic polymorphisms of ALDH2, an isozyme of ALDH, and the plasma pharmacokinetics (PK) of VACV, ACV and CMMG in subjects with end-stage renal disease on hemodialysis.

ELIGIBILITY:
Inclusion criteria:

* Japanese subjects with chronic renal failure undergoing hemodialysis regularly three times a week for at least 12 weeks prior to the start of the study.

Exclusion criteria:

* Subjects with current alcohol dependence.
* Subjects with gastrointestinal dysfunction that may affect drug absorption.
* Subjects who have received an organ transplant (However, subjects with a corneal transplant or any other organ transplant that may not affect the objectives of the study will be eligible for inclusion in this study).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2005-07; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
- The pharmacokinetic parameters for VACV, ACV and CMMG - Relationship between ALDH2 genotypes and the pharmacokinetics of VACV, ACV and CMMG in blood

SECONDARY OUTCOMES:
- Change in blood ACV and CMMG concentrations after a 4-hour hemodialysis session - Safety (adverse events occurring during the study, clinical laboratory tests)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline